CLINICAL TRIAL: NCT07153588
Title: Awareness and Perception of Glaucoma Among Patients Attending Ophthalmology OPD in a Tertiary Care Hospital: A Prospective Study.
Brief Title: Awareness and Perception of Glaucoma Among Patients Attending Ophthalmology OPD in a Tertiary Care Hospital.
Status: Completed | Type: Observational
Sponsor: Bacha Khan Medical College (Other)
Responsible Party: Principal Investigator, Malik Shayan Ali Khan, Doctor, Bacha Khan Medical College
Other Study IDs: Ref no. 771/BKMC
Record Dates: First submitted 2025-08-25; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Level of awareness — This study uses a structured, interviewer-assisted questionnaire as the main intervention. The questionnaire is designed to assess patients' awareness and perception of glaucoma. It includes four sections:
  Sociodemographic information (age, gender, education, occupation, residence, family history)
  Ocular history (diagnosis of glaucoma, history of eye disease, surgery, or previous eye checkups)
  Awareness of glaucoma (understanding of risk factors, symptoms, prevention, and treatment options)
  Perceptions and attitudes (beliefs about curability, reversibility of vision loss, and willingness for screening and education).
  For illiterate participants, trained research staff will administer the questionnaire verbally without influencing responses. The data collection method distinguishes this intervention from treatment-based studies, as it focuses on knowledge assessment and perception analysis rather than a medical or surgical procedure.

SUMMARY:
Glaucoma is often called the "silent thief of vision" because it can slowly damage the optic nerve and cause permanent blindness if it is not found and treated early. Many people are not aware of glaucoma, its risk factors, or the importance of regular eye checkups.

This study is being conducted at the Ophthalmology Outpatient Department of Mardan Medical Complex, a large tertiary care hospital in Pakistan. The aim is to find out how much patients know and understand about glaucoma, and what beliefs or misconceptions they may have.

A total of 379 patients between the ages of 18 and 80 years will be asked to complete a simple questionnaire. The questions cover background information, eye history, knowledge about glaucoma, and attitudes toward screening and treatment. For patients who cannot read, trained staff will help them complete the questionnaire.

The information from this study will help doctors and health policy makers design better educational programs, improve public awareness, and encourage early eye screening. This can reduce the risk of irreversible vision loss caused by glaucoma

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness worldwide and is often described as the "silent thief of vision." Because it progresses slowly and early symptoms are often missed, many patients only seek medical care after significant vision has already been lost. Lack of awareness and misconceptions about glaucoma are major barriers to early diagnosis and treatment, particularly in low- and middle-income countries.

This study is designed to measure the awareness and perception of glaucoma among patients attending the Ophthalmology Outpatient Department of a tertiary care hospital in Mardan, Pakistan. Using a structured questionnaire, researchers will collect information on four domains:

Sociodemographic details (age, gender, education, occupation, residence, and family history of glaucoma)

Ocular history (previous eye disease, surgery, or diagnosis of glaucoma)

Awareness of glaucoma (understanding of risk factors, symptoms, and treatment)

Perceptions and attitudes (beliefs about curability, reversibility of vision loss, and willingness to undergo screening or learn more).

A total of 379 participants will be included, and assistance will be provided for patients who cannot read or write to ensure accurate responses. Statistical analysis will be used to identify patterns and factors associated with higher or lower awareness levels.

The findings are expected to highlight critical knowledge gaps, common misconceptions, and areas where targeted educational efforts are most needed. By identifying who is most at risk of poor awareness, this study will provide evidence for developing effective public health interventions, awareness campaigns, and screening programs. Ultimately, the results aim to support earlier diagnosis and better management of glaucoma, reducing preventable vision loss in the community.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18 and 80 years of age attending the Ophthalmology Outpatient Department (new or follow-up cases).
* Patients with ocular conditions, including diagnosed glaucoma and other eye pathologies.

Exclusion Criteria:

* Patients with cognitive impairment or mental illness that limits their ability to understand or respond to the questionnaire.
* Patients with ocular malignancy or active ocular bleeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients aged 18 to 80 years who attend the Ophthalmology Outpatient Department (OPD) at Mardan Medical Complex, a tertiary care teaching hospital in Khyber Pakhtunkhwa, Pakistan. Both new and follow-up patients are included, regardless of whether they have glaucoma or another eye condition.
  Participants come from a variety of backgrounds, with many residing in rural areas and a large proportion having limited or no formal education. Patients with diagnosed glaucoma, those with other ocular problems such as cataract or refractive errors, and individuals with systemic conditions like diabetes or hypertension are all eligible.
  Patients unable to provide informed responses due to cognitive impairment, mental illness, ocular malignancy, or active ocular bleeding are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Level of Awareness about Glaucoma | At the time of questionnaire completion (baseline, single visit)
  Proportion of participants who demonstrate correct perception of glaucoma, defined as identifying it as a disease associated with increased intraocular pressure and risk of irreversible vision loss.

SECONDARY OUTCOMES:
Perception of Glaucoma and Its Curability | (Baseline, single visit)
  Percentage of participants who believe glaucoma is curable, reversible, or leads to permanent blindness.

CONTACTS AND LOCATIONS:
Locations (1):
- Mardan Medical Comlex, Mardan, Mardan, KPK, Pakistan